CLINICAL TRIAL: NCT07405814
Title: An International, Randomized, Double-Blind, Placebo-Controlled Clinical Trial On The Effect Of Artisterol On Metabolic And Vascular Risk Factors In Individuals With Suboptimal Cholesterol Levels
Brief Title: Clinical Trial On The Effect Of Artisterol On Risk Factors In Individuals With Suboptimal Cholesterol Levels
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zentiva, k.s. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CINARL1118125
Record Dates: First submitted 2025-09-29; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Hyperlipoproteinemia
MeSH Terms: conditions — Hyperlipoproteinemias | interventions — Thiamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Artisterol (Experimental)
  Interventions: Dietary Supplement: investigational product containing phytosterol, artichoke extract and thiamin
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: investigational product containing phytosterol, artichoke extract and thiamin — subjects will take the investigational product once daily
  Arms: Artisterol
Other: Placebo — matching placebo administration
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn if Artisterol works to lower LDL cholesterol and other metabolic and vascular risk factors in adults. The main questions it aims to answer are:

• Does Artisterol lower low-density lipoprotein cholesterol (LDL-C) levels in participants and by how much? Researchers will compare Artisterol to a placebo (a look-alike substance that contains no drug) to see if Artisterol works to lower LDL cholesterol.

Participants will:

* Take drug Artisterol or a placebo every day for 3 months
* Visit the clinic once every 6 weeks for checkups and tests
* Keep a diary of their Artisterol intake and physical activity

DETAILED DESCRIPTION:
This study is designed to test if a new food supplement, called Artisterol, can help lower cholesterol levels in adults. High cholesterol is a common health issue that increases the risk of heart disease by causing fatty buildups in the arteries. This research will provide evidence on the supplement's ability to decrease "bad" cholesterol (LDL-C) and will also check its safety and how well it is tolerated.

The supplement being tested, Artisterol, contains natural active ingredients including plant sterols, artichoke extract, and vitamin B1. The study will compare its effects to a placebo, which is a substance that looks and tastes identical but has no active ingredients.

This is a "randomized, double-blind, placebo-controlled" study. This means that participants will be randomly assigned, like flipping a coin, to one of two groups: one group will receive Artisterol, and the other will receive the placebo. The study is "double-blind," which means neither the participants nor the study doctors will know who is receiving the active supplement and who is receiving the placebo until the study is complete. This method helps prevent bias and ensures the results are reliable.

Who can participate? The study is looking for at least 106 adults, both men and women, between the ages of 18 and 70. Participants should have mildly high LDL-C ("bad" cholesterol) levels, specifically between 115 and 160 mg/dL, and not be currently taking medication to lower their cholesterol. Participants must be willing to follow the study's procedures and dietary recommendations. Individuals who are pregnant or breastfeeding, have certain severe medical conditions, or are allergic to the supplement's ingredients are not eligible to participate.

What does participation involve? The study involves a treatment period of 12 weeks. Participants will be asked to take one sachet of their assigned supplement (Artisterol or placebo) orally each day.

Participation includes:

* A screening visit (V1) to confirm eligibility, which involves signing an informed consent form, a physical exam, and blood tests.
* A baseline visit (V2) to be officially enrolled and receive the 12-week supply of the study supplement.
* Two follow-up clinic visits at Week 6 (V3) and Week 12 (V4) for physical check-ups and further blood sample collections.

The main goal of the study is to measure the change in participants' LDL-C levels from the beginning of the study to the end at Week 12. Researchers will compare the results between the group taking Artisterol and the group taking the placebo to see if the supplement is effective. The study will also look at changes in other blood fats (like total cholesterol and triglycerides) and markers for liver and metabolic health. Throughout the study, participants' health and safety will be carefully monitored.

ELIGIBILITY:
Inclusion Criteria:

1. Female or male, 18-70 years old.
2. Subjects with mild hypercholesterolemia previously untreated (LDL-C levels between 115 and 160 mg/dL. Note that the upper limit can be extended to 190 mg/dL in case of subject refusing another treatment or intolerant to statins or other lipid lowering therapies. If previously treated, washout of 3 months is required.
3. Written informed consent has been obtained during screening visit prior to any study specific procedure.
4. Subject must understand the informed consent form and other study documents and are willing and able to comply with scheduled visits and requirements of the study protocol, including study specific Dietary Recommendations .
5. Subject must be healthy or stabilized based on medical history and physical examination.
6. Females of childbearing potential must have a negative pregnancy test at screening and agree to use a highly effective form of birth control while on study (from Screening through final study visit).

Exclusion Criteria:

1. Pregnant or lactating females
2. Specific feeding regimens if not stabilized between screening and baseline, especially those in conflict with study specific Dietary Recommendation.
3. Subjects receiving therapies and medications, that may affect lipid levels. If used in the past, washout of 3 months is required.
4. Subjects who have a medical condition or history that limits the subject to adhere to the protocol schedule and requirements:

   1. Known or suspected allergy to the content of investigational product
   2. Previous or ongoing severe medical or laboratory abnormality (acute or chronic) which, in the judgement of the investigator, would make the subject inappropriate for entry into the study
   3. Subjects under a long-term treatment. Subjects stable for 30 days are allowed in the study
   4. Subjects with a history of acute myocardial infarction (AMI) or severe cardiac conditions
   5. Subjects with a history of alcoholism, drug and subjects with severe psychotic disorders (stable anti-depressive treatments are allowed)
   6. Subjects unable to understand and follow the study procedures
5. Subjects who are currently participate in another interventional clinical study. Historical participation in a clinical study is allowed with 3 months of washout period (after last IMP dose).
6. Subject with family or hierarchical relationships with the research team members at clinical site.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2026-02-02 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Absolute mean change in Low-density-lipoprotein-cholesterol levels / mg/dl | from baseline to Week 12
  The absolute mean change in fasting Low-Density Lipoprotein Cholesterol (LDL-C) levels from baseline to Week 12.Units: mg/dL,

SECONDARY OUTCOMES:
Absolute mean changes in Total Cholesterol, High-Density-Lipoprotein-Cholesterol, Non-High-Density-Lipoprotein-Cholesterol and Triglycerides / mg/dl | from baseline to Week 12
  Absolute mean change in Total Cholesterol levels from baseline to Week 12. Units: mg/dl
Absolute mean change in Apolipoprotein-B level / mg/dl | from baseline to Week 12
  Absolute mean change in Apolipoprotein B (ApoB) levels from baseline to Week 12. ApoB reflects the total number of atherogenic particles. Units: mg/dl
Absolute mean changes in glutamat-oxalacetat-transaminase, glutamate pyruvate transaminase, and gamma-glutamyl transferase levels | from baseline to Week 12
  Absolute mean change in Aspartate Aminotransferase (also known as Glutamate Oxaloacetate Transaminase or GOT) levels from baseline to Week 12 / U/l Absolute mean change in Alanine Aminotransferase (also known as Glutamate Pyruvate Transaminase or GPT) levels from baseline to Week 12 / U/l Absolute mean change in Gamma-Glutamyl Transferase levels from baseline to Week 12 / U/l
Mean change in Fasting plasma glucose levels Unit: mg/dl | from baseline to Week 12
  Absolute mean change in fasting plasma glucose levels from baseline to Week 12 / mg/dl
Number of Participants With Clinically Significant Physical Examination Abnormalities. Unit: participants | Week 12
  The number of participants who have physical examination findings assessed as "Abnormal, Clinically Significant" by the investigator at the end of the study. Assessment includes evaluation of general appearance, cardiovascular, respiratory, and gastrointestinal systems.
Incidence of Concomitant Medication Use. Unit: participants | Baseline through Week 12
  The number of participants experiencing at least one Adverse Event (AE) during the treatment period. An AE is defined as any untoward medical occurrence in a participant which does not necessarily have a causal relationship with the treatment.
Incidence of Adverse Events (TEAEs) Unit: participants | Baseline through Week 12
  The number of participants experiencing at least one Adverse Event (AE) during the treatment period. An AE is defined as any untoward medical occurrence in a participant which does not necessarily have a causal relationship with the treatment.